CLINICAL TRIAL: NCT00855582
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multinational Study to Evaluate the Efficacy and Safety of Tadalafil 2.5 and 5 mg Once Daily Dosing for 12 Weeks for the Treatment of Erectile Dysfunction and Signs and Symptoms of Benign Prostatic Hyperplasia in Men With Both Erectile Dysfunction and Benign Prostatic Hyperplasia
Brief Title: A Study in the Treatment of Erectile Dysfunction and Benign Prostate Hyperplasia
Acronym: COMORBID©
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11667; H6D-MC-LVHR (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Erectile Dysfunction; Benign Prostatic Hyperplasia
Keywords: Erectile Dysfunction; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tadalafil 2.5 mg (Experimental)
  Interventions: Drug: Tadalafil
- Tadalafil 5 mg (Experimental)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — tablet once daily by mouth for 12 weeks.
  Other Names: Cialis; LY450190
  Arms: Tadalafil 2.5 mg; Tadalafil 5 mg
Drug: Placebo — Matching 2.5 or 5 mg placebo tablet once daily by mouth for 12 weeks.
  Arms: Placebo

SUMMARY:
Study LVHR is a Phase 3 study which will examine the efficacy and safety of tadalafil 2.5 and 5 mg once daily versus placebo for the treatment of erectile dysfunction (ED) and signs and symptoms of benign prostatic hyperplasia (BPH) in men with both ED and signs and symptoms of BPH.

ELIGIBILITY:
Inclusion Criteria:

* Have BPH Lower Urinary Tract Symptoms (LUTS) based on the disease diagnostic criteria at 1st screening.
* Have a history of ED based on the disease diagnostic criteria at 1st screening.
* Have LUTS with a Total International Prostate Symptom Score (IPSS) greater than or equal to 13 at 2nd screening.
* Have bladder outlet obstruction as defined by a Peak Urine Flow Rate (Qmax) of greater than or equal to 4 to less than or equal to 15 milliliter (mL)/second (sec) (from a prevoid total bladder volume as assessed by ultrasound of greater than or equal to 150 to less than or equal to 550 mL and a minimum voided volume of 125 mL) at 2nd screening.
* Make at least 4 sexual intercourse attempts during the 4-weeks after 2nd screening as recorded in the Sexual Encounter Profile (SEP) diary.
* Are sexually active with an adult female partner, and expect to remain sexually active with the same adult female partner for the duration of the study.
* Agree not to use any other approved or experimental BPH, overactive bladder (OAB), or ED treatments as indicated in the protocol at any time during the study.
* Have not taken treatments indicated in the protocol prior to the 2nd screening.

Exclusion Criteria:

* Current treatment with nitrates.
* Prostate-specific antigen (PSA) greater than 10.0 nanogram (ng)/mL at 1st screening.
* PSA greater than or equal to 4.0 to less than or equal to 10.0 ng/mL at 1st screening if prostate malignancy has not been ruled out to the satisfaction of a urologist.
* Clinical evidence of prostate cancer.
* Bladder postvoid residual volume (PVR) greater than or equal to 300 mL by ultrasound determination at 1st screening.
* History or clinical evidence of certain pelvic, bladder, urinary tract, or urinary retention conditions described in the protocol.
* Lower urinary tract instrumentation (including prostate biopsy) within 30 days of 1st screening.
* Clinical evidence of severe hepatic impairment at 1st screening.
* Current neurologic disease or condition associated with neurogenic bladder (for example, Parkinson's disease or multiple sclerosis).
* History of significant renal insufficiency as defined by the protocol.
* History of ED caused by other primary sexual disorders including premature ejaculation or ED caused by untreated endocrine disease.
* Presence of penile deformity judged by the investigator to be clinically significant.
* History of certain cardiac or cardiovascular conditions described in the protocol.
* History of resuscitated cardiac arrest.
* Current treatment with certain medications described in the protocol.
* Scheduled or planned surgery (or any procedure requiring general, spinal, or epidural anesthesia) during the course of the study.
* History of significant central nervous system injuries (including stroke or spinal cord injury) within 6 months of 1st screening.
* Glycosylated hemoglobin (HbA1c) greater than 9% at 1st screening.
* Prior treatment with phosphodiesterase type 5 (PDE5) inhibitors judged by the investigator to be ineffective. However, if the investigator judges that a subject's lack of response to as-needed PDE5 inhibitors is the result of inadequate coordination between dosing and sexual activity with a treatment, the subject may be enrolled.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarzana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Englewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Urbana, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmond, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mountlake Terrace, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint John, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carpentras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Rappenau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holzminden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempen
- Greece (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trieste
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Joya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
- Portugal (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amadora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don

REFERENCES:
- [Derived] Vlachopoulos C, Oelke M, Maggi M, Mulhall JP, Rosenberg MT, Brock GB, Esler A, Buttner H. Impact of cardiovascular risk factors and related comorbid conditions and medical therapy reported at baseline on the treatment response to tadalafil 5 mg once-daily in men with lower urinary tract symptoms associated with benign prostatic hyperplasia: an integrated analysis of four randomised, double-blind, placebo-controlled, clinical trials. Int J Clin Pract. 2015 Dec;69(12):1496-507. doi: 10.1111/ijcp.12722. Epub 2015 Aug 24. PMID 26299520
- [Derived] Porst H, Gacci M, Buttner H, Henneges C, Boess F. Tadalafil once daily in men with erectile dysfunction: an integrated analysis of data obtained from 1913 patients from six randomized, double-blind, placebo-controlled, clinical studies. Eur Urol. 2014 Feb;65(2):455-64. doi: 10.1016/j.eururo.2013.09.037. Epub 2013 Oct 2. PMID 24119319

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is a 4-week washout during Screening in order to assess symptoms and uroflowmetry data in the absence of therapy. After the screening/washout period, subjects began a 4-week single-blind, placebo lead-in period to assess treatment and study procedure compliance and to establish baseline levels.
Groups:
- Tadalafil 2.5 mg: 2.5 mg tablet once daily by mouth for 12 weeks.
- Tadalafil 5 mg: 5 mg tablet once daily by mouth for 12 weeks.
- Placebo: Matching placebo tablet once daily by mouth for 12 weeks.
Period: Overall Study
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Started | 198 | 208 | 200
Completed | 172 | 184 | 170
Not Completed | 26 | 24 | 30
Not completed — Adverse Event | 2 | 6 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 8
Not completed — Lost to Follow-up | 1 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 6 | 2 | 6
Not completed — Entry Criteria Not Met | 8 | 6 | 3
Not completed — Withdrawal by Subject | 7 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo | Total
Number analyzed (Participants) | 198 | 208 | 200 | 606
Age Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.56) | 62.5 (8.43) | 62.9 (8.23) | 62.6 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 198 | 208 | 200 | 606
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 31 | 30 | 94
  Not Hispanic or Latino | 165 | 177 | 170 | 512
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 6 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 8 | 23
  White | 181 | 194 | 190 | 565
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 17 | 24 | 21 | 62
  Portugal | 8 | 3 | 6 | 17
  United States | 71 | 71 | 68 | 210
  Mexico | 27 | 27 | 22 | 76
  Canada | 22 | 23 | 26 | 71
  Greece | 7 | 9 | 9 | 25
  Russian Federation | 21 | 29 | 25 | 75
  Germany | 10 | 12 | 9 | 31
  Italy | 15 | 10 | 14 | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kg/m² | 27.7 (3.86) | 28.0 (4.18) | 28.6 (4.8) | 28.1 (4.3)
Lower Urinary Tract Symptoms (LUTS) Severity [Number; unit: participants] — The total IPSS is obtained by combining the scores of the responses to component questions 1 through 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  participants
    Moderate (IPSS <20) | 123 | 124 | 122 | 369
    Severe (IPSS ≥20) | 74 | 84 | 78 | 236
    Unknown | 1 | 0 | 0 | 1
Peak Urine Flow Rate (Qmax) [Number; unit: participants]
  <10 mL/sec | 96 | 87 | 99 | 282
  10-15 mL/sec | 73 | 83 | 66 | 222
  >15mL/sec | 21 | 16 | 16 | 53
  Unknown | 8 | 22 | 19 | 49
Postvoid Residual Volume (PRV) [Mean (Standard Deviation); unit: mL] | 53.0 (51.24) | 51.1 (60.91) | 55.5 (60.46) | 53.2 (57.72)
Erectile Dysfunction (ED) - Etiology [Number; unit: participants]
  Psychogenic | 13 | 15 | 12 | 40
  Organic | 65 | 70 | 85 | 220
  Mixed | 76 | 83 | 63 | 222
  Unknown | 44 | 40 | 40 | 124
ED - Severity [Number; unit: participants] — Self-reported erectile function over the past 4 weeks. Scores range from 0 (low or no erectile function) to 5 (high erectile function) on 6 questions (1-5, 15 of the IIEF). Total Erectile Function Domain scores range from 0 to 30; lower numerical scores represent greater severity of erectile dysfunction.
  participants
    Mild (IIEF EF Domain 17-30) | 104 | 99 | 93 | 296
    Moderate (IIEF EF Domain 11-16) | 46 | 54 | 49 | 149
    Severe (IIEF EF Domain 1-10) | 48 | 55 | 58 | 161
ED - Duration [Number; unit: participants]
  <1 year | 12 | 20 | 19 | 51
  ≥1 year | 186 | 188 | 181 | 555

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 12 Endpoint (5 mg)
Description: The total IPSS is obtained by combining the scores of the responses to component questions 1 through 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tadalafil 5 mg: Tablet once daily by mouth for 12 weeks.
Arm/Group | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 206 | 194
units on a scale | -6.1 (0.43) | -3.8 (0.45)
Statistical Analysis 1: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed using a Dunnett-Bonferroni gatekeeping procedure for multiple hypothesis testing. The pre-specified alpha level of 0.0271 was used; ANCOVA model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction; Median Difference (Final Values) = -2.3, Standard Error of Mean 0.58

2. Primary Outcome: Change From Baseline in International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score at Week 12 Endpoint (5 mg)
Description: Self-reported erectile function over the past 4 weeks. Questions 1-5 were scored from 0-5, and Question 15 from 1 to 5. Erectile Function Domain scores range from 1 to 30; lower numerical scores represent greater severity of erectile dysfunction. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 203 | 190
units on a scale | 6.5 (0.49) | 1.8 (0.51)
Statistical Analysis 1: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.7, Standard Error of Mean 0.66

3. Primary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 12 Endpoint (2.5 mg)
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tadalafil 2.5 mg: Tablet once daily by mouth for 12 weeks.
Arm/Group | Tadalafil 2.5 mg | Placebo
Number analyzed (Participants) | 191 | 194
units on a scale | -4.6 (0.44) | -3.8 (0.45)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.181, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, Standard Error of Mean 0.59

4. Primary Outcome: Change From Baseline in International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score at Week 12 Endpoint (2.5 mg)
Description: as for outcome 2
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Placebo
Number analyzed (Participants) | 190 | 190
units on a scale | 5.2 (0.5) | 1.8 (0.51)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.4, Standard Error of Mean 0.67

5. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 3 at Week 12 Endpoint (5 mg)
Description: Assessed as the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3, "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of Yes responses per the number of sexual attempts for a participant during a study period. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of Yes responses
Arm/Group | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 199 | 187
percentage of Yes responses | 31.7 (2.07) | 12.0 (2.14)
Statistical Analysis 1: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed using a Dunnett-Bonferroni gatekeeping procedure for multiple hypothesis testing. The pre-specified alpha level of 0.0228 was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 19.7, Standard Error of Mean 2.80

6. Secondary Outcome: Change From Baseline in Benign Prostatic Hyperplasia (BPH) Impact Index (BII) at Week 12 Endpoint (5 mg)
Description: The BII is a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores range from 0 to 13; higher scores represent increased perceived impact of benign prostatic hyperplasia-lower urinary tract symptoms on overall health. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 203 | 190
units on scale | -2.1 (0.19) | -1.2 (0.20)
Statistical Analysis 1: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.26

7. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 3 at Week 12 Endpoint (2.5 mg)
Description: as for outcome 5
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of yes responses
Arm/Group | Tadalafil 2.5 mg | Placebo
Number analyzed (Participants) | 185 | 187
percentage of yes responses | 24.6 (2.11) | 12.0 (2.14)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed using a Dunnett-Bonferroni gatekeeping procedure for multiple hypothesis testing. Based on the results of prior tests under this procedure, the statistical significance of this hypothesis was not assessed; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.5, Standard Error of Mean 2.85

8. Secondary Outcome: Change From Baseline in BPH Impact Index (BII) at Week 12 Endpoint (2.5 mg)
Description: as for outcome 6
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Placebo
Number analyzed (Participants) | 190 | 190
units on a scale | -1.6 (0.20) | -1.2 (0.20)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.156, ANCOVA — [p-value comment as in outcome 7, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, Standard Error of Mean 0.26

9. Secondary Outcome: Change From Baseline in Modified IPSS (mIPSS) at Week 2 Endpoint
Description: The Modified IPSS is the total IPSS collected at 2 weeks post-baseline. The total IPSS is obtained by combining the scores of the responses to component questions 1 through 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from ANCOVA. The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 148 | 160 | 162
units on a scale | -2.8 (0.39) | -4.0 (0.38) | -2.2 (0.38)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.226, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, Standard Error of Mean 0.50

10. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) at Week 4 and Week 8 Endpoint
Description: as for outcome 1
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 198 | 208 | 200
units on a scale
  Week 4 Change (n=184, 197, 183) | -3.4 (0.39) | -5.5 (0.38) | -2.6 (0.40)
  Week 8 Change (n=174, 192, 178) | -4.5 (0.43) | -5.8 (0.41) | -3.8 (0.43)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.121, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons. P-value is for change from Baseline at Week 4. Change= Week 4 minus Baseline; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.169, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons. P-value is for change from Baseline at Week 8. Change= Week 8 minus Baseline; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, Standard Error of Mean 0.57
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.9, Standard Error of Mean 0.52
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, Standard Error of Mean 0.56

11. Secondary Outcome: Change From Baseline in International Index of Erectile Function - Erectile Function (IIEF-EF) Domain at Week 4 and Week 8 Endpoint
Description: as for outcome 2
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 198 | 208 | 200
units on a scale
  Week 4 Change (n=186, 197, 183) | 4.2 (0.44) | 6.1 (0.43) | 1.0 (0.45)
  Week 8 Change (n=176, 192, 178) | 4.9 (0.49) | 6.6 (0.48) | 1.8 (0.52)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.1, Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.1, Standard Error of Mean 0.71
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.0, Standard Error of Mean 0.59
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.8, Standard Error of Mean 0.71

12. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 3 at Week 4 and Week 8 Endpoint
Description: as for outcome 5
Time Frame: Baseline, 4 weeks, 8 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of yes responses
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 198 | 208 | 200
percentage of yes responses
  Week 4 Change (n=180, 190, 180) | 22.3 (2.31) | 30.7 (2.27) | 6.2 (2.35)
  Week 8 Change (n=172, 187, 171) | 22.9 (2.16) | 31.7 (2.11) | 10.9 (2.21)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.1, Standard Error of Mean 3.1
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.0, Standard Error of Mean 3.0
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 24.5, Standard Error of Mean 3.1
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 20.9, Standard Error of Mean 2.9

13. Secondary Outcome: Change From Baseline in BPH Impact Index (BII) at Week 4 and 8 Endpoint
Description: as for outcome 6
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 198 | 208 | 200
units on a scale
  Week 4 Change (n=186, 197, 183) | -1.0 (0.17) | -1.5 (0.16) | -0.7 (0.17)
  Week 8 Change (n=175, 192, 177) | -1.4 (0.18) | -1.8 (0.17) | -1.2 (0.18)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.215, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.325, ANOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 10, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.23

14. Secondary Outcome: Change From Baseline in International Prostate Symptom Score Voiding (Obstructive) Subscore at Week 12 Endpoint
Description: IPSS obstructive subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. The obstructive subscore ranges from 0 to 20 with a higher score representing greater obstruction. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 191 | 206 | 194
units on a scale | -2.7 (0.28) | -3.6 (0.28) | -2.2 (0.29)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.230, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, Standard Error of Mean 0.37

15. Secondary Outcome: Change From Baseline in International Prostate Symptom Score Storage (Irritative) Subscore at Week 12 Endpoint
Description: IPSS irritative subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. The irritative subscore ranges from 0 to 15 with a higher score representing more irritative symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 192 | 206 | 194
units on a scale | -1.9 (0.2) | -2.5 (0.19) | -1.6 (0.20)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.191, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.3

16. Secondary Outcome: Change From Baseline in International Prostate Symptom Score Nocturia Question at Week 12
Description: The IPSS Nocturia question (Question 7) measures the number of times needed to get up at night to urinate. Scores range from 0 (none) to 5 (5 or more times). Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 192 | 206 | 194
units on a scale | -0.5 (0.08) | -0.6 (0.07) | -0.5 (0.08)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.763, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0, Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.075, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, Standard Error of Mean 0.1

17. Secondary Outcome: Change From Baseline in International Prostate Symptom Score Quality of Life (QoL) at Week 12 Endpoint
Description: Assessment of quality of life (QoL) by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible). Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 192 | 205 | 194
units on a scale | -0.9 (0.10) | -1.0 (0.10) | -0.8 (0.11)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.384, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.082, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.1

18. Secondary Outcome: Change From Baseline in International Index of Erectile Function - Overall Satisfaction Domain at Week 12 Endpoint
Description: Self-reported overall satisfaction over the past 4 weeks. Calculated as the sum of IIEF Questions 13 and 14. Each question is scored from 1 through 5, with a possible total score of 2 through 10. Higher scores represent greater satisfaction. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 190 | 203 | 190
units on a scale | 1.8 (0.16) | 2.4 (0.16) | 0.5 (0.16)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.9, Standard Error of Mean 0.2

19. Secondary Outcome: Change From Baseline in International Index of Erectile Function - Intercourse Satisfaction Domain at Week 12 Endpoint
Description: Self-reported intercourse satisfaction over the past 4 weeks. Calculated as the sum of IIEF Questions 6, 7 and 8. Each question is scored from 0 through 5 with a possible total score of 0 through 15. Higher score represent greater satisfaction. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 190 | 203 | 190
units on a scale | 1.6 (0.23) | 2.0 (0.22) | 0.2 (0.23)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.9, Standard Error of Mean 0.3

20. Secondary Outcome: Change From Baseline in International Index of Erectile Function Question 3 at Week 12 Endpoint
Description: IIEF Question 3 asks how often a subject was able to penetrate his partner over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 190 | 203 | 190
units on a scale | 0.9 (0.10) | 1.1 (0.10) | 0.2 (0.10)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7, Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.1

21. Secondary Outcome: Change From Baseline in International Index of Erectile Function Question 4 at Week 12 Endpoint
Description: IIEF Question 4 asks whether how often a subject was able to maintain an erection after penetration over the past 4 weeks. Scores range from 0 (did not attempt intercourse) to 5 (almost always or always). Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 190 | 203 | 190
units on a scale | 0.9 (0.11) | 1.3 (0.10) | 0.4 (0.11)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5, Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.1

22. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 2 at Week 12 Endpoint
Description: Assessed as the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2, "Were you able to insert your penis into your partner's vagina?" Data are presented as the mean percentage of yes responses per the number of sexual attempts for a participant during a study period. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of yes responses
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 185 | 199 | 187
percentage of yes responses | 21.4 (1.82) | 25.1 (1.78) | 9.3 (1.84)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.1, Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 15.8, Standard Error of Mean 2.4

23. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 4 at Week 12 Endpoint
Description: Assessed as the mean change from baseline in the percentage of Yes responses to the SEP diary Question 4, "Were you satisfied with the hardness of your erection?" Data are presented as the mean percentage of yes responses per the number of sexual attempts for a participant during a study period. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of yes responses
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 185 | 199 | 187
percentage of yes responses | 26.6 (2.48) | 39.4 (2.46) | 9.6 (2.61)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.9, Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 29.7, Standard Error of Mean 3.6

24. Secondary Outcome: Change From Baseline in Yes Responses to Sexual Encounter Profile (SEP) Diary Question 5
Description: Assessed as the mean change from baseline in the percentage of Yes responses to the SEP diary Question 5, "Were you satisfied overall with this sexual experience?" Data are presented as the mean percentage of yes responses per the number of sexual attempts for a participant during a study period. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, baseline covariate, baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: percentage of yes responses
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 185 | 199 | 187
percentage of yes responses | 23.7 (2.49) | 38.2 (2.48) | 9.9 (2.63)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.8, Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 28.4, Standard Error of Mean 3.6

25. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at Week 12 Endpoint
Description: A scale that measures the patient's perception of urinary symptoms at endpoint compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). The data are presented as the number of participants in each of the seven categories: very much better (1); much better (2); a little better (3); no change (4); a little worse (5); much worse (6); very much worse (7).
Time Frame: 12 weeks
Population: Participants started study medication, and had non-missing data.
Measure: Number; unit: participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 185 | 197 | 185
participants
  Very Much Worse | 0 | 0 | 1
  Much Worse | 3 | 2 | 4
  A Little Worse | 12 | 3 | 13
  No Change | 34 | 34 | 61
  A Little Better | 66 | 79 | 63
  Much Better | 57 | 60 | 37
  Very Much Better | 13 | 19 | 6
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; The Cochran-Mantel-Haenszel test was adjusted for baseline LUTS severity
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; The Cochran-Mantel-Haenszel test was adjusted for baseline LUTS severity

26. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) at Week 12 Endpoint
Description: A scale that measures clinician's rating of the total change in the patient's urinary symptoms at endpoint compared with the start of treatment. Scores range from 1 (very much better) to 7 (very much worse).The data are presented as the number of participants in each of the seven categories: very much better (1); much better (2); a little better (3); no change (4); a little worse (5); much worse (6); very much worse (7).
Time Frame: 12 weeks
Population: Participants started study medication, and had non-missing data.
Measure: Number; unit: participants
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 181 | 197 | 184
participants
  Very Much Worse | 0 | 0 | 1
  Much Worse | 2 | 1 | 4
  A Little Worse | 8 | 2 | 9
  No Change | 41 | 42 | 64
  A Little Better | 67 | 60 | 58
  Much Better | 56 | 78 | 45
  Very Much Better | 7 | 14 | 3
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; The Cochran-Mantel-Haenszel test was adjusted for baseline LUTS severity
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons; The Cochran-Mantel-Haenszel test was adjusted for baseline LUTS severity

27. Secondary Outcome: Erectile Function General Assessment Questionnaire (EF-GAQ)
Description: The EF-GAQ consisted of two questions: (1) Has the treatment you have been taking during this study improved your erections? and (2) If yes, has the treatment improved your ability to engage in sexual activity? Each question has a Yes/No response.
Time Frame: 12 weeks
Population: Participants started study medication, and had non-missing data.
Measure: Number; unit: participants with yes response
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 184 | 196 | 185
participants with yes response
  Question 1 | 135 | 155 | 74
  Question 2 | 126 | 146 | 67
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons. P-value is for Question 1; Logistic regression model includes terms for treatment group, region and centered-baseline IIEF EF Domain score
Statistical Analysis 2: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons. P-value is for Question 2; Logistic regression model includes terms for treatment group, region and centered-baseline IIEF EF Domain score
Statistical Analysis 3: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 27, analysis 1]; Logistic regression model includes terms for treatment group, region and centered-baseline IIEF EF Domain score
Statistical Analysis 4: Comparison: Tadalafil 5 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 27, analysis 2]; Logistic regression model includes terms for treatment group, region and centered-baseline IIEF EF Domain score

28. Secondary Outcome: Change From Baseline in Uroflowmetry Parameters - Peak Urine Flow Rate (Qmax) at Week 12 Endpoint
Description: Qmax is defined as the peak urine flow rate (measured in milliliters per second [mL/sec] using standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 milliliters (mL) and the voided volume (Vcomp) was >= 125 mL.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 157 | 160 | 143
mL/sec | 1.7 (4.45) | 1.6 (4.15) | 1.2 (4.52)
Statistical Analysis 1: Comparison: Tadalafil 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.027, Ranked ANOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Tadalafil 5 mg vs Placebo; Test type: Superiority or Other; p = 0.186, Ranked ANOVA — Statistical significance was assessed at an alpha level of 0.05 with no adjustments for multiple comparisons

29. Secondary Outcome: Change From Baseline in Uroflowmetry Parameters - Mean Urine Flow Rate (Qmean) at Week 12 Endpoint
Description: Qmean is defined as the average urine flow rate (measured in milliliters per second [mL/second] using standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 milliliters (mL) and the voided volume (Vcomp) was >= 125 mL.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 157 | 161 | 143
mL/sec | 1.0 (2.65) | 0.9 (2.92) | 0.6 (2.6)

30. Secondary Outcome: Change From Baseline in Uroflowmetry Parameters - Voided Volume (Vcomp) at Week 12 Endpoint
Description: Vcomp is defined as the volume of urine voided (measures in mL using a standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 milliliters (mL) and the voided volume (Vcomp) was >= 125 mL.
Time Frame: Baseline, 12 weeks
Population: Participants with non-missing baseline value and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Number analyzed (Participants) | 157 | 161 | 143
mL | 18.5 (113.9) | 13.3 (92.75) | 11.4 (91.84)

ADVERSE EVENTS:
Arm/Group | Tadalafil 2.5 mg | Tadalafil 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/198 | 1/208 | 1/200
Other Adverse Events (participants affected / at risk) | 50/198 | 56/208 | 38/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 2.5 mg (N=198) | Tadalafil 5 mg (N=208) | Placebo (N=200)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — This event resulted in death.
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 2.5 mg (N=198) | Tadalafil 5 mg (N=208) | Placebo (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 1 (1) | 5 (5)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (5) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Scan myocardial perfusion abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2)
Drooling (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 12 (12) | 6 (6)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Terminal dribbling (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
P-values for the peak urine flow rate outcome were corrected in this record after an error was identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days